CLINICAL TRIAL: NCT01760005
Title: A Phase II/III Multicenter Randomized, Double-Blind, Placebo-Controlled Platform Trial of Potential Disease Modifying Therapies Utilizing Biomarker, Cognitive, and Clinical Endpoints in Dominantly Inherited Alzheimer's Disease
Brief Title: Dominantly Inherited Alzheimer Network Trial: An Opportunity to Prevent Dementia. A Study of Potential Disease Modifying Treatments in Individuals at Risk for or With a Type of Early Onset Alzheimer's Disease Caused by a Genetic Mutation. Master Protocol DIAN-TU-001
Acronym: DIAN-TU
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eli Lilly and Company (Industry); Hoffmann-La Roche (Industry); Alzheimer's Association (Other); National Institute on Aging (NIA) (NIH); Avid Radiopharmaceuticals (Industry); Accelerating Medicines Partnership (AMP) (Other); Eisai Inc. (Industry); Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIAN-TU-001 (Master); The Alzheimer's Association (Other Grant/Funding Number: DIAN TTU-12-243040); U01AG042791 (NIH); 2013-000307-17 (EudraCT Number); R01AG046179 (NIH); REec-2014-0817 (Registry Identifier: Spanish Clinical Studies Registry); The Alzheimer's Association (Other Grant/Funding Number: DIAN-TU Tau-15-347219); GHR Foundation (Other Grant/Funding Number: File 4401); Alzheimer's Association (Other: HDE 18S84914); The Alzheimer's Association (Other Grant/Funding Number: DIAN-TU NG-16-434362); R56AG053267 (NIH); U01AG059798 (NIH); R01AG053267 (NIH)
Record Dates: First submitted 2012-12-26; First posted 2013-01-03 (Estimated); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Alzheimers Disease; Dementia; Alzheimers Disease, Familial
Keywords: Alzheimer's; Alzheimer's Disease; Dementia; Mutation; Genetic Mutation; Dominantly Inherited Alzheimer's Disease; Dominantly Inherited Alzheimer Network; Autosomal Dominant Alzheimer's Disease; Early Onset Alzheimer's Disease; DIAN; DIAN-TU; DIAN TU; DIAD
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — gantenerumab; solanezumab; lecanemab

STUDY DESIGN:
Intervention Model Description: Interventional with a non-interventional run-in component (Future interventions to be added)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: One arm is Open-label as noted in the arm descriptions
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Gantenerumab (Experimental): This arm completed and is closed.
  Interventions: Drug: Gantenerumab
- Solanezumab (Experimental): This arm completed and is closed.
  Interventions: Drug: Solanezumab
- Matching placebo (Gantenerumab) (Placebo Comparator): This arm completed and is closed.
  Interventions: Drug: Matching Placebo (Gantenerumab)
- Matching Placebo (Solanezumab) (Placebo Comparator): This arm completed and is closed.
  Interventions: Drug: Matching Placebo (Solanezumab)
- Cognitive Run-in (No Intervention): This arm is completed and closed.
- Gantenerumab Open Label Extension (Active Comparator): Subcutaneously every 4 weeks at escalating doses. This arm is completed and closed.
  Interventions: Drug: Gantenerumab
- E2814 plus lecanemab (Experimental): Symptomatic Population (Cohort 1)
  At Week 0, participants will receive open-label lecanemab administered intravenously for the full treatment period.
  At Week 24, participants randomized to E2814 will receive intravenously in a blinded fashion for the remainder of their treatment period.
  Asymptomatic Population (Cohort 2)
  At Week 0, participants randomized to E2814 will receive intravenously in a blinded fashion for the full treatment period.
  At Week 52, all participants will initiate open-label lecanemab administered intravenously for the remainder of their treatment period.
  Interventions: Drug: E2814; Drug: Lecanemab
- Matching placebo (E2814) plus lecanemab (Experimental): Symptomatic Population (Cohort 1)
  At Week 0, participants will receive open-label lecanemab administered intravenously for the full treatment period.
  At Week 24, participants randomized to E2814 placebo will receive placebo intravenously in a blinded fashion for the remainder of their treatment period.
  Asymptomatic Population (Cohort 2)
  At Week 0, participants randomized to E2814 placebo will receive placebo intravenously in a blinded fashion for the full treatment period.
  At Week 52, all participants will initiate open-label lecanemab administered intravenously for the remainder of their treatment period.
  Interventions: Drug: Lecanemab; Drug: Matching Placebo (E2814)

INTERVENTIONS:
Drug: Gantenerumab — Subcutaneously every 4 weeks at escalating doses
  Other Names: RO4909832
  Arms: Gantenerumab
Drug: Solanezumab — Intravenous infusion every 4 weeks at escalating doses
  Other Names: LY2062430
  Arms: Solanezumab
Drug: Matching Placebo (Gantenerumab) — Subcutaneous injection of placebo every 4 weeks
  Arms: Matching placebo (Gantenerumab)
Drug: Matching Placebo (Solanezumab) — Intravenous infusion of placebo every 4 weeks
  Arms: Matching Placebo (Solanezumab)
Drug: Gantenerumab — Open-label administered Subcutaneously every 4 weeks at escalating doses
  Other Names: RO4909832
  Arms: Gantenerumab Open Label Extension
Drug: E2814 — Administered intravenously in a blinded fashion
  Arms: E2814 plus lecanemab
Drug: Lecanemab — Administered intravenously
  Other Names: BAN2401
  Arms: E2814 plus lecanemab; Matching placebo (E2814) plus lecanemab
Drug: Matching Placebo (E2814) — Placebo administered intravenously in a blinded fashion.
  Arms: Matching placebo (E2814) plus lecanemab

SUMMARY:
The purpose of this study is to assess the safety, tolerability, biomarker, cognitive and clinical efficacy of investigational products in participants with an Alzheimer's disease-causing mutation by determining if treatment with the study drug slows the rate of progression of cognitive/clinical impairment or improves disease-related biomarkers.

DETAILED DESCRIPTION:
This study will recruit participants from the Dominantly Inherited Alzheimer Network (DIAN) observational study, a multicenter international study supported by the National Institutes of Health (Grant Number U01-AG032438; RJ Bateman), Dominantly Inherited Alzheimer Network Trial Units (DIAN-TU) sites, DIAN-TU partner sites, DIAN Expanded Registry (DIAN-EXR), and families identified by the sites. As part of the DIAN-TU-001 protocol, participants undergo longitudinal assessments that include clinical assessment, cognitive testing, magnetic resonance imaging (MRI) and amyloid and tau positron emission tomography (PET) imaging, and analysis of blood and cerebrospinal fluid (CSF).

Participants in DIAN are recruited from families that have at least one member who has been identified as having a mutation linked to dominantly inherited Alzheimer's disease (DIAD). The mutations in presenilin 1 (PSEN1), presenilin 2 (PSEN2) and amyloid precursor protein (APP) that are associated with dominantly inherited Alzheimer's disease have very high penetrance (near 100%). This study enrolls individuals who are either known to have a disease-causing mutation or who are at risk for such a mutation (the descendant or sibling of a proband with a known mutation) and unaware of their genetic status. Because the age at onset of cognitive changes is relatively consistent within each family and with each mutation, an age at onset is determined for each affected parent or mutation as part of the DIAN Observational (DIAN-OBS) study protocol. This study will enroll participants who are either asymptomatic and are within a specific window of time of expected age at onset for their family and/or mutation or who have symptoms of mild Alzheimer's disease.

The ability to identify individuals destined to develop Alzheimer's disease (AD) and predict the age of onset with a high degree of confidence provides a unique opportunity to assess the efficacy of therapies at asymptomatic and very early stages of dementia. Families with known disease-causing mutations are extremely rare and are geographically dispersed throughout the world. These constraints necessitate a specialized study design. Many of the participants in this study will not yet have any cognitive symptoms of AD; they will be "asymptomatic" carriers of mutations that cause dominantly inherited Alzheimer's disease and would be expected to perform normally on standard cognitive and functional testing. Imaging and fluid biomarkers will be used to demonstrate that the treatment compounds have engaged their therapeutic targets. A set of cognitive measures designed to assess the very earliest and most subtle cognitive changes will be collected. Additionally, because many at-risk individuals decide not to know whether they have the disease-associated mutation or not, when allowable in individual drug arms, some of the at-risk individuals enrolled in this study will not have the disease-causing mutations; they will be "mutation negative". It is important to enroll these participants to avoid coercion (e.g., potential participants may be pressured into genetic testing to learn their genetic status in order to be eligible for the trial) unless the drug-specific design includes open-label treatment. These mutation negative individuals will be assigned to the placebo group and data will be used to determine normal ranges of outcome measures. Participants and site study staff will remain blinded as to these individuals' active or placebo group assignment and mutation status. Thus, the study will be double-blinded for placebo and for mutation status, except for mutation positive participants who are aware of their genetic status. There may be exceptional circumstances when required by local regulation or health authorities where enrollment may be restricted to mutation carriers only, but such mandates will be thoroughly documented and agreed upon by the governing regulatory agency and sponsor.

This is an adaptive platform-based study. Several different therapies (each referred to as a study drug arm) will be tested in order to increase the likelihood that an effective treatment will be discovered. The compounds are selected for this trial based on mechanism of action and available data on efficacy and safety profile. The study design includes a pooled placebo group (referred to as the mutation positive placebos) which may be shared by study drug arms. Mutation positive participants will be assigned to a study drug arm and subsequently randomized within that arm to the active drug to placebo ratio specified in each drug-specific appendix. When included in individual drug arms, mutation negative participants will all receive placebo treatment. Participants and study staff will not be blinded as to which study drug arm each participant has been assigned; they will be blinded as to whether participants have been randomized to active drug or placebo.

Biomarker, cognitive, and/or clinical endpoints will be specified for each study drug arm. Biomarker data will be analyzed for pre-specified endpoints consistent with the drug's mechanism of action and other AD biomarker outcomes.

Interim analyses of the imaging or fluid biomarker endpoint will assess safety and whether each study drug engages its biological targets. The clinical and cognitive assessments are designed to assess subtle cognitive changes that may be detectable before the onset of dementia as well as cognitive and clinical decline in symptomatic groups.

After the last participant in a study drug arm completes the 4-year treatment period, participants in that study drug arm may be eligible to receive active study drug in an open-label extension period.

A cognitive run-in (CRI) period was implemented to allow for enrollment during periods when study drug arms are not randomizing. This enables the DIAN-TU platform to have continuous enrollment during periods before or in-between drug arm randomization.

The CRI period of cognitive, clinical, and imaging data collection was designed as part of the platform study to utilize the time in between enrollment of study drug arms. The CRI period will enhance study enrollment by identifying eligible participants and engaging them with the cognitive assessments and can reduce practice effects by allowing participants to habituate to the testing process. The CRI further provides important baseline and run-in data that adds control data to the platform and informs about the effects of tested drugs. The data collected in the CRI period will be used for analysis in the respective drug arm under which participants are randomized and treated.

Solanezumab and gantenerumab double blind treatment arms: Primary Completion Date= Nov 2019 and Study Completion= March 2020 (NCT04623242)

Gantenerumab open-label extension was discontinued based on findings from an interim efficacy analysis and the status of the drug program. Primary Completion Date= October 6, 2023; Study final completed visit= November 13, 2023 (NCT06424236)

E2814 treatment arm enrollment complete: Primary Completion Date= April 2028 and Study Completion= July 2028 (NCT05269394)

ELIGIBILITY:
Inclusion Criteria:

* Between 18-80 years of age
* Individuals who know they have an Alzheimer's disease-causing mutation or are unaware of their genetic status and have dominantly inherited Alzheimer's disease (DIAD) mutation in their family.
* Are within -15 to + 10 years of the predicted or actual age of cognitive symptom onset. For Cognitive Run-In (CRI): includes participants who are younger than 15 years prior to the expected age of cognitive symptom onset, in addition to those 15 years younger and no more than 10 years older than expected or actual age of cognitive symptom onset.
* Cognitively normal or with mild cognitive impairment or mild dementia, Clinical Dementia Rating (CDR) of 0-1 (inclusive)
* Fluency in DIAN-TU trial approved language and evidence of adequate premorbid intellectual functioning
* Able to undergo Magnetic Resonance Imaging (MRI), Lumbar Puncture (LP), Positron Emission Tomography (PET), and complete all study related testing and evaluations.
* For women of childbearing potential, if partner is not sterilized, subject must agree to use effective contraceptive measures (hormonal contraception, intra-uterine device, sexual abstinence, barrier method with spermicide).
* Adequate visual and auditory abilities to perform all aspects of the cognitive and functional assessments.
* Has a Study Partner who in the investigator's judgment is able to provide accurate information as to the subject's cognitive and functional abilities, who agrees to provide information at the study visits which require informant input for scale completion.

Exclusion Criteria:

* History or presence of brain MRI scans indicative of any other significant abnormality
* Alcohol or drug dependence currently or within the past 1 year
* Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, or foreign metal objects in the eyes, skin or body which would preclude MRI scan.
* History or presence of clinically significant cardiovascular disease, hepatic/renal disorders, infectious disease or immune disorder, or metabolic/endocrine disorders
* Anticoagulants except low dose (≤ 325 mg) aspirin.
* Have been exposed to a monoclonal antibody targeting beta amyloid peptide within the past six months.
* History of cancer within the last 5 years, except basal cell carcinoma, non-squamous skin carcinoma, prostate cancer or carcinoma in situ with no significant progression over the past 2 years.
* Positive urine or serum pregnancy test or plans or desires to become pregnant during the course of the trial.
* Subjects unable to complete all study related testing, including implanted metal that cannot be removed for MRI scanning, required anticoagulation and pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2012-12 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Assess cognitive efficacy in individuals with mutations causing dominantly inherited AD as measured by the change from baseline in the DIAN-Multivariate Cognitive Endpoint (DIAN-MCE) | Baseline and Weeks 52, 104, 156, and 208
  The DIAN-Multivariate Cognitive Endpoint (DIAN-MCE) consists of 4 cognitive measures: Wechsler Memory Scale-Revised Logical Memory Delayed Recall Test, Wechsler Adult Intelligence Sale Digit Symbol Substitution Test (WAIS), International Shopping List Task (ISLT), Mini-Mental State Examination (MMSE)

CONTACTS AND LOCATIONS:
Overall Officials: Randall J Bateman, MD, Study Director — Washington University School of Medicine
Locations (38):
- United States (12):
  - University of Alabama in Birmingham, Birmingham, Alabama
  - University of California San Diego Medical Center, La Jolla, California
  - USC Keck School of Medicine, Los Angeles, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Washington University in St. Louis, St Louis, Missouri
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Butler Hospital, Providence, Rhode Island
  - Kerwin Medical Center, Dallas, Texas
  - University of Washington, Seattle, Washington
- Instituto de Investigaciones Neurologicas Raul Carrea, FLENI, Ciudad Autonoma de Buenos Aire, Argentina
- Australia (3):
  - Neuroscience Research Australia, Randwick, New South Wales
  - Mental Health Research Institute, Melbourne, Victoria
  - The McCuster Foundation of Alzheimer's Disease Research, Nedlands, Western Australia
- Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, Brazil
- Canada (4):
  - UBC Hospital, Vancouver, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - McGill Center for Studies in Aging, Verdun, Quebec
  - CHU de Quebec - Hôpital de l' Enfant Jésus, Québec
- Grupo de Neurociencias Sede de la Universidad de Antioquia, Medellín, Colombia
- France (5):
  - CHU de Toulouse - Hôpital Purpan, Toulouse, Haute Garonne
  - Hopital Roger Salengro - CHU Lille, Lille, Nord
  - Groupe Hospitalier Pitie-Salpetriere, Paris, Paris
  - Hopital Neurologique Pierre Wertheimer, Bron, Rhone
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen, Seine Maritime
- Germany (2):
  - Universitaetsklinikum Tubingen, Tübingen, Baden-Wurttemberg
  - LMU-Campus Grosshadern, Munich, Bavaria
- St Vincent's University Hospital, Dublin, Dublin, Ireland
- Italy (2):
  - IRCCS Centro San Giovanni di Dio Fatebenefratelli, Brescia
  - Azienda Ospedaliera Universitaria Careggi, Florence
- Japan (2):
  - Niigata University Medical & Dental Hospital, Niigata, Niigata
  - University of Tokyo Hospital, Bunkyō City, Tokyo-To
- Brain Research Center, Amsterdam, Netherlands
- University of Puerto Rico, School of Medicine, San Juan, Puerto Rico, Puerto Rico
- Hospital Clínic I Provincial de Barcelona, Barcelona, Barcelona, Spain
- The National Hospital for Neurology and Neurosurgery, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to DIAN-TU trial data will follow the DIAN-TU data access policy, which complies with the guidelines established by the Collaboration for Alzheimer's Prevention [CAP REF].

REFERENCES:
- [Background] Bateman RJ, Xiong C, Benzinger TL, Fagan AM, Goate A, Fox NC, Marcus DS, Cairns NJ, Xie X, Blazey TM, Holtzman DM, Santacruz A, Buckles V, Oliver A, Moulder K, Aisen PS, Ghetti B, Klunk WE, McDade E, Martins RN, Masters CL, Mayeux R, Ringman JM, Rossor MN, Schofield PR, Sperling RA, Salloway S, Morris JC; Dominantly Inherited Alzheimer Network. Clinical and biomarker changes in dominantly inherited Alzheimer's disease. N Engl J Med. 2012 Aug 30;367(9):795-804. doi: 10.1056/NEJMoa1202753. Epub 2012 Jul 11. PMID 22784036
- [Background] Farlow M, Arnold SE, van Dyck CH, Aisen PS, Snider BJ, Porsteinsson AP, Friedrich S, Dean RA, Gonzales C, Sethuraman G, DeMattos RB, Mohs R, Paul SM, Siemers ER. Safety and biomarker effects of solanezumab in patients with Alzheimer's disease. Alzheimers Dement. 2012 Jul;8(4):261-71. doi: 10.1016/j.jalz.2011.09.224. Epub 2012 Jun 5. PMID 22672770
- [Background] Bateman RJ, Benzinger TL, Berry S, Clifford DB, Duggan C, Fagan AM, Fanning K, Farlow MR, Hassenstab J, McDade EM, Mills S, Paumier K, Quintana M, Salloway SP, Santacruz A, Schneider LS, Wang G, Xiong C; DIAN-TU Pharma Consortium for the Dominantly Inherited Alzheimer Network. The DIAN-TU Next Generation Alzheimer's prevention trial: Adaptive design and disease progression model. Alzheimers Dement. 2017 Jan;13(1):8-19. doi: 10.1016/j.jalz.2016.07.005. Epub 2016 Aug 29. PMID 27583651
- [Background] Mills SM, Mallmann J, Santacruz AM, Fuqua A, Carril M, Aisen PS, Althage MC, Belyew S, Benzinger TL, Brooks WS, Buckles VD, Cairns NJ, Clifford D, Danek A, Fagan AM, Farlow M, Fox N, Ghetti B, Goate AM, Heinrichs D, Hornbeck R, Jack C, Jucker M, Klunk WE, Marcus DS, Martins RN, Masters CM, Mayeux R, McDade E, Morris JC, Oliver A, Ringman JM, Rossor MN, Salloway S, Schofield PR, Snider J, Snyder P, Sperling RA, Stewart C, Thomas RG, Xiong C, Bateman RJ. Preclinical trials in autosomal dominant AD: implementation of the DIAN-TU trial. Rev Neurol (Paris). 2013 Oct;169(10):737-43. doi: 10.1016/j.neurol.2013.07.017. Epub 2013 Sep 6. PMID 24016464
- [Background] Wang G, Berry S, Xiong C, Hassenstab J, Quintana M, McDade EM, Delmar P, Vestrucci M, Sethuraman G, Bateman RJ; Dominantly Inherited Alzheimer Network Trials Unit. A novel cognitive disease progression model for clinical trials in autosomal-dominant Alzheimer's disease. Stat Med. 2018 Sep 20;37(21):3047-3055. doi: 10.1002/sim.7811. Epub 2018 May 14. PMID 29761523
- [Background] Weninger S, Carrillo MC, Dunn B, Aisen PS, Bateman RJ, Kotz JD, Langbaum JB, Mills SL, Reiman EM, Sperling R, Santacruz AM, Tariot PN, Welsh-Bohmer KA. Collaboration for Alzheimer's Prevention: Principles to guide data and sample sharing in preclinical Alzheimer's disease trials. Alzheimers Dement. 2016 May;12(5):631-2. doi: 10.1016/j.jalz.2016.04.001. No abstract available. PMID 27157073
- [Background] Grill JD, Bateman RJ, Buckles V, Oliver A, Morris JC, Masters CL, Klunk WE, Ringman JM; Dominantly Inherited Alzheimer's Network. A survey of attitudes toward clinical trials and genetic disclosure in autosomal dominant Alzheimer's disease. Alzheimers Res Ther. 2015 Jul 22;7(1):50. doi: 10.1186/s13195-015-0135-0. eCollection 2015. PMID 26203303
- [Background] McDade E, Bateman RJ. Stop Alzheimer's before it starts. Nature. 2017 Jul 12;547(7662):153-155. doi: 10.1038/547153a. No abstract available. PMID 28703214
- [Background] McDade E, Wang G, Gordon BA, Hassenstab J, Benzinger TLS, Buckles V, Fagan AM, Holtzman DM, Cairns NJ, Goate AM, Marcus DS, Morris JC, Paumier K, Xiong C, Allegri R, Berman SB, Klunk W, Noble J, Ringman J, Ghetti B, Farlow M, Sperling RA, Chhatwal J, Salloway S, Graff-Radford NR, Schofield PR, Masters C, Rossor MN, Fox NC, Levin J, Jucker M, Bateman RJ; Dominantly Inherited Alzheimer Network. Longitudinal cognitive and biomarker changes in dominantly inherited Alzheimer disease. Neurology. 2018 Oct 2;91(14):e1295-e1306. doi: 10.1212/WNL.0000000000006277. Epub 2018 Sep 14. PMID 30217935
- [Background] Ryman DC, Acosta-Baena N, Aisen PS, Bird T, Danek A, Fox NC, Goate A, Frommelt P, Ghetti B, Langbaum JB, Lopera F, Martins R, Masters CL, Mayeux RP, McDade E, Moreno S, Reiman EM, Ringman JM, Salloway S, Schofield PR, Sperling R, Tariot PN, Xiong C, Morris JC, Bateman RJ; Dominantly Inherited Alzheimer Network. Symptom onset in autosomal dominant Alzheimer disease: a systematic review and meta-analysis. Neurology. 2014 Jul 15;83(3):253-60. doi: 10.1212/WNL.0000000000000596. Epub 2014 Jun 13. PMID 24928124
- [Background] Weng H, Bateman R, Morris JC, Xiong C. Validity and power of minimization algorithm in longitudinal analysis of clinical trials. Biostat Epidemiol. 2017;1(1):59-77. doi: 10.1080/24709360.2017.1331822. Epub 2017 Jun 13. PMID 29250611
- [Derived] Bateman RJ, Li Y, McDade EM, Llibre-Guerra JJ, Clifford DB, Atri A, Mills SL, Santacruz AM, Wang G, Supnet C, Benzinger TLS, Gordon BA, Ibanez L, Klein G, Baudler M, Doody RS, Delmar P, Kerchner GA, Bittner T, Wojtowicz J, Bonni A, Fontoura P, Hofmann C, Kulic L, Hassenstab J, Aschenbrenner AJ, Perrin RJ, Cruchaga C, Renton AE, Xiong C, Goate AA, Morris JC, Holtzman DM, Snider BJ, Mummery C, Brooks WS, Wallon D, Berman SB, Roberson E, Masters CL, Galasko DR, Jayadev S, Sanchez-Valle R, Pariente J, Kinsella J, van Dyck CH, Gauthier S, Hsiung GR, Masellis M, Dubois B, Honig LS, Jack CR, Daniels A, Aguillon D, Allegri R, Chhatwal J, Day G, Fox NC, Huey E, Ikeuchi T, Jucker M, Lee JH, Levey AI, Levin J, Lopera F, Roh J, Rosa-Neto P, Schofield PR; Dominantly Inherited Alzheimer's Disease-Trials Unit. Safety and efficacy of long-term gantenerumab treatment in dominantly inherited Alzheimer's disease: an open-label extension of the phase 2/3 multicentre, randomised, double-blind, placebo-controlled platform DIAN-TU trial. Lancet Neurol. 2025 Apr;24(4):316-330. doi: 10.1016/S1474-4422(25)00024-9. PMID 40120616
- [Derived] Bateman RJ, Li Y, McDade EM, Llibre-Guerra JJ, Clifford DB, Atri A, Mills SL, Santacruz AM, Wang G, Supnet C, Benzinger TLS, Gordon BA, Ibanez L, Klein G, Baudler M, Doody RS, Delmar P, Kerchner GA, Bittner T, Wojtowicz J, Bonni A, Fontoura P, Hofmann C, Kulic L, Hassenstab J, Aschenbrenner AJ, Perrin RJ, Cruchaga C, Renton AE, Xiong C, Goate AA, Morris JC, Holtzman DM, Snider BJ, Mummery C, Brooks WS, Wallon D, Berman SB, Roberson E, Masters CL, Galasko DR, Jayadev S, Sanchez-Valle R, Pariente J, Kinsella J, van Dyck CH, Gauthier S, Robin Hsiung GY, Masellis M, Dubois B, Honig LS, Jack CR, Daniels A, Aguillon D, Allegri R, Chhatwal J, Day G, Fox N, Huey E, Ikeuchi T, Jucker M, Lee JH, Levey AI, Levin J, Lopera F, Roh J, Rosa-Neto P, Schofield PR; Dominantly Inherited Alzheimer's Disease-Trials Unit. Safety and efficacy of long-term gantenerumab treatment in dominantly inherited Alzheimer's disease: an open label extension of the phase 2/3 multicentre, randomised, double-blind, placebo-controlled platform DIAN-TU Trial. medRxiv [Preprint]. 2025 Jan 29:2024.10.29.24316289. doi: 10.1101/2024.10.29.24316289. PMID 39974075
- [Derived] Chen CD, McCullough A, Gordon B, Joseph-Mathurin N, Flores S, McKay NS, Hobbs DA, Hornbeck R, Fagan AM, Cruchaga C, Goate AM, Perrin RJ, Wang G, Li Y, Shi X, Xiong C, Pontecorvo MJ, Klein G, Su Y, Klunk WE, Jack C, Koeppe R, Snider BJ, Berman SB, Roberson ED, Brosch J, Surti G, Jimenez-Velazquez IZ, Galasko D, Honig LS, Brooks WS, Clarnette R, Wallon D, Dubois B, Pariente J, Pasquier F, Sanchez-Valle R, Shcherbinin S, Higgins I, Tunali I, Masters CL, van Dyck CH, Masellis M, Hsiung R, Gauthier S, Salloway S, Clifford DB, Mills S, Supnet-Bell C, McDade E, Bateman RJ, Benzinger TLS; DIAN-TU Study Team. Longitudinal head-to-head comparison of 11C-PiB and 18F-florbetapir PET in a Phase 2/3 clinical trial of anti-amyloid-beta monoclonal antibodies in dominantly inherited Alzheimer's disease. Eur J Nucl Med Mol Imaging. 2023 Jul;50(9):2669-2682. doi: 10.1007/s00259-023-06209-0. Epub 2023 Apr 5. PMID 37017737
- See also: Expanded registry — http://www.dianexr.org/